CLINICAL TRIAL: NCT04428879
Title: Phase I Sustained-Release Topotecan Episcleral Plaque (Chemoplaque) for Retinoblastoma
Brief Title: Topotecan Episcleral Plaque for Treatment of Retinoblastoma
Acronym: STEP-RB
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Brenda Gallie, Head, Retinoblastoma Program, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1000064742
Record Dates: First submitted 2020-06-04; First posted 2020-06-11 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-10

CONDITIONS: Retinoblastoma
Keywords: Retinal Neoplasms; Neoplasms; Eye Neoplasms; Eye Diseases, Hereditary; Eye Diseases; Retinal Diseases; Topotecan
MeSH Terms: conditions — Retinoblastoma; Retinal Neoplasms; Neoplasms; Eye Neoplasms; Eye Diseases, Hereditary; Eye Diseases; Retinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Phase I single arm trial (Experimental)
  Interventions: Drug: Topotecan Episcleral Plaque

INTERVENTIONS:
Drug: Topotecan Episcleral Plaque — Sustained Release Episcleral Topotecan Plaques (Chemoplaques) are glued to bare, dry sclera of the eye under conjunctiva and Tenon's capsule. A rolling six dose interpatient escalation schema will be employed. Chemoplaques with 0.6 mg and 0.9 mg of topotecan HCl formulation are available. Patients will receive 1 or 2 Chemoplaques per eye, to deliver 5 escalating doses: 0.6, 0.9, 1.2 [2x0.6], 1.5 [0.6+0.9] or 1.8 [2x0.9] mg. The prescribed dose will escalate or de-escalate by 0.3 mg at each level, and no patient will receive more than 1.8 mg of topotecan hydrochloride due to the physical limitations if the devices available. The planned removal is 42 days ± 7, unless dose limiting toxicity is observed, in which case the plaque is removed as soon as possible. The observation period for the purposes of dose-escalation will be 63 days (i.e. 21 days following Chemoplaque removal on day 42).
  Other Names: Episcleral Topotecan; Transscleral Topotecan; Sustained Release Episcleral Topotecan; Chemoplaque

SUMMARY:
This single site, single-arm, non-randomized, dose escalation phase I toxicity clinical trial will assess primarily the safety and secondarily the efficacy of episcleral topotecan in patients with active de novo or residual or recurrent intraocular retinoblastoma in at least one eye following completion of first-line therapy.

DETAILED DESCRIPTION:
Retinoblastoma is the most common pediatric malignant intraocular tumour and originates from the retina. Treatment of eyes with advanced intraocular retinoblastoma remains a challenge. The historic standard of care for patients with unilateral disease is enucleation and for those with bilateral disease, a variety of modalities have been tried. These include radiation therapy, systemic chemotherapy, periocular administration of chemotherapy, selective intra-arterial chemotherapy, and intravitreal chemotherapy. Unfortunately, all of these modalities are associated with significant morbidity and investigators are looking for new ways to treat these patients either with novel directed drug delivery methods or with new less toxic agents. This study will evaluate the safety and efficacy of topotecan delivered directly to the eye using a novel sustained-release topotecan episcleral plaque (also referred to as a Chemoplaque) in patients with active residual or recurrent intraocular retinoblastoma in at least one eye following completion of first-line therapy. The study intervention involves the insertion and removal of the Chemoplaque, examinations under anaesthesia (EUAs), visits to clinic to monitor for adverse events throughout, and post plaque removal toxicity evaluation. EUAs, clinic visits and laboratory tests are standard of care for retinoblastoma patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age. Participants must be <18 years of age.
2. Diagnosis and Treatment. Participants must have: (i) active residual or recurrent intraocular retinoblastoma following completion of first-line therapy (chemotherapy, systemic or intra-arterial, focal therapy or brachytherapy), or (ii) unilateral Group B, C, D or cT1b, cT2 retinoblastoma at diagnosis with no previous treatment.
3. One eye will be the Study Eye. When participants have two eyes with retinoblastoma, the eye with worst disease or best vision potential will be designated the Study Eye. There will only be one eye per child treated in this Phase I study, since treatment of two eyes would double the systemic dose of drug. The Non-study eye will be treated by standard of care, with only focal therapy during the Study Period, if required.
4. Disease status. Study eye must have vision potential and no clinical features suggestive of high risk of extraocular extension.
5. Performance status. Lansky play score ≥ 50 if <16 years of age; Karnofsky performance scale of ≥ 50 if ≥16 years of age (Appendix I)
6. Organ function:

   1. Adequate bone marrow function and platelet count
   2. Adequate renal function
   3. Adequate liver function
7. Pregnancy prevention. Females of reproductive potential must agree to the use of highly effective contraception during study participation and for an additional 40 days after the end of the Chemoplaque administration
8. Informed consent. All participants and/or their parents or legally authorized representatives must have the ability to understand and the willingness to sign a written informed consent. Assent, where appropriate, will also be obtained.

Exclusion Criteria:

1. Disease status. Participants known to have any of the following are excluded:

   1. clinical or EUA evidence of extraocular extension
   2. known metastatic disease status and intercurrent illness
   3. existing clinical and neuroimaging showing suspicion of, or definitive,
2. Allergy. Participants with reported allergy to topotecan, camptothecin or derivatives thereof.
3. Concomitant treatment. Participants may not receive chemotherapy or other focal retinoblastoma therapy or any other investigational agent within 3 weeks of the placement and removal of the Chemoplaque, nor while the Chemoplaque is in situ.
4. Uncontrolled intercurrent illness. Participants with known uncontrolled intercurrent illness that, in the investigator's opinion, would put the participant at undue risk or limit compliance with the study requirements.
5. Febrile illness. Participants with clinically significant febrile illness (as determined by the investigator) within one week prior to initiation of protocol therapy.
6. Pregnancy and lactation. Females of reproductive potential must have a negative serum pregnancy test within 72 hours prior to initiation of protocol therapy. Due to the unknown but potential risk for adverse events (AEs) in nursing infants secondary to treatment of the mother with the study agents, breastfeeding must be discontinued if the mother is treated on study.
7. Compliance. Any condition of diagnosis that could in the opinion of the Principal Investigator or delegate interfere with the participant's ability to comply with the study instruction, might confound the interpretation of the study results, or put the participant at risk.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2020-06-16 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-03 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose and Recommended Phase 2 Dose of topotecan hydrochloride administered as a Chemoplaque to pediatric patients with active Retinoblastoma. | 9 weeks
  Inter-Patient Escalation in the rolling six phase 1 trial design will determine Maximum Tolerated Dose and Recommended Phase 2 Dose. Dose level assignment is based on the number of participants currently enrolled in the cohort, the number of dose limiting toxicities observed, and the number of participants at risk for developing a dose limiting toxicity (i.e., participants enrolled but who are not yet assessable for toxicity).

SECONDARY OUTCOMES:
Tumor response to the Chemoplaque as secondary therapy in eye(s) with active retinoblastoma after completion of primary standard of care treatment. | 9 weeks
  Tumor response will be characterized as (i) complete regression, (ii) very good (iii) partial regression, (iv) partial regression, (v) stable disease or (vi) progressive disease determined by evaluating number of tumour sites, appearance and tumour size.

CONTACTS AND LOCATIONS:
Overall Officials: Brenda Gallie, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No